CLINICAL TRIAL: NCT00003725
Title: Phase III Randomized Study of a Single Adjunctive Instillation of Intravesical AD 32 (N-Trifluoroacetyladriamycin-14-valerate) Versus No Adjunctive Therapy Immediately Following Transurethral Resection in Patients With Multiple Superficial (Ta/T1) Bladder Tumors
Brief Title: Surgery With or Without Chemotherapy in Treating Patients With Newly Diagnosed or Recurrent Bladder Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Anthra Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000066837; ANTHRA-A9601
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-05

CONDITIONS: Bladder Cancer
Keywords: stage 0 bladder cancer; stage I bladder cancer; recurrent bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — valrubicin

INTERVENTIONS:
Drug: valrubicin
Procedure: conventional surgery

SUMMARY:
RATIONALE: Transurethral resection is a less invasive type of surgery for bladder cancer and may have fewer side effects and improve recovery. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether transurethral resection plus AD 32 is more effective than transurethral resection alone for bladder cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of transurethral resection surgery followed by AD 32 with that of transurethral resection alone in treating patients who have newly diagnosed or recurrent bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy of adjuvant AD 32 following complete transurethral resection versus transurethral resection alone in patients with newly diagnosed or recurrent superficial transitional cell carcinoma of the bladder. II. Assess the toxicity of AD 32 in these patients.

OUTLINE: This is an open label, randomized, multicenter study. Patients are randomized to receive surgery with AD 32 or surgery alone. Arm I: Patients undergo surgery to remove bladder tumors. AD 32 is administered by catheter into the bladder within 2-24 hours after surgery. Patients must hold the AD 32 liquid in the bladder for 90 minutes. Arm II: Patients undergo only surgery to remove bladder tumors. Patients with T1 or Tis disease may receive BCG therapy once weekly for 6 weeks, followed by 6 weeks of rest. Patients are followed every 3 months for 2 years.

PROJECTED ACCRUAL: This study will accrue approximately 300 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed stage 0 (Ta), stage I, or recurrent superficial transitional cell carcinoma of the bladder Must have at least 2 papillary appearing bladder tumors by cystoscopic examination Patients with recurrent disease must have no history of Tis tumor

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: Not specified Hematopoietic: WBC greater than 4000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) SGOT no greater than 2 times ULN Renal: Creatinine no greater than 2 times ULN Other: Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biological response modifiers for bladder cancer Chemotherapy: No prior or concurrent chemotherapy for bladder cancer No prior AD 32 therapy for bladder cancer Endocrine therapy: Not specified Radiotherapy: No prior or concurrent radiotherapy Surgery: At least 9 months since any complete transurethral resection of the bladder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 1996-12

CONTACTS AND LOCATIONS:
Overall Officials: Peter R. Carroll, MD, Study Chair — University of California, San Francisco
Locations (53):
- United States (51):
  - Urology Associates, Birmingham, Alabama
  - Urology Associates, Ltd., Phoenix, Arizona
  - University of California San Diego Cancer Center, La Jolla, California
  - San Diego Urology Center, La Mesa, California
  - Hillcrest Urological Medical Group, San Diego, California
  - San Diego Urology Center, San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Santa Monica Urologic Medical Group, Santa Monica, California
  - Western Urological Associates, Van Nuys, California
  - Urology Specialists, P.C., Waterbury, Connecticut
  - George Washington University Hospital, Washington D.C., District of Columbia
  - Atlantic Urological Associates, Daytona Beach, Florida
  - University of Florida - Gainesville, Gainesville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Urology Care - South, Miami, Florida
  - Urology Health Center, New Port Richey, Florida
  - Office of Ira W. Klimberg, Ocala, Florida
  - Urology Treatment Center, Sarasota, Florida
  - Georgia Urology, Atlanta, Georgia
  - Affliated Urology, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Clinic of Urologic Wellness, Lexington, Kentucky
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Cambridge Urological Associates, Inc., Cambridge, Massachusetts
  - Michigan Institute of Urology, Detroit, Michigan
  - Mississippi Urology Clinic, P.A., Jackson, Mississippi
  - Urology Center, Omaha, Nebraska
  - Sheldon Freedman Ltd., Las Vegas, Nevada
  - Desert Urology, North Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Office of John Byrne, New Rochelle, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Wake Urological Associates, Raleigh, North Carolina
  - Department of Urology and Urologic Oncology, Columbus, Ohio
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Urology Clinic, P.C., Portland, Oregon
  - Office of Jeffrey K. Cohen, Pittsburgh, Pennsylvania
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - Vanderbilt Cancer Center, Nashville, Tennessee
  - Urology Associates of North Texas, Arlington, Texas
  - Baylor College of Medicine, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Sentara Cancer Center, Norfolk, Virginia
  - Virginia Urology Center, Richmond, Virginia
  - Office of Ronald G. Anderson, Tacoma, Washington
  - West Virginia University Hospitals, Morgantown, West Virginia
- Canada (2):
  - Ottawa General Hospital, Ottawa, Ontario
  - Toronto General Hospital, Toronto, Ontario